CLINICAL TRIAL: NCT01311674
Title: Hepatitis B Virus (HBV) Antibody (Anti-HBs) Booster Program for the Production of Hepatitis B Immune Globulin (HBIG)
Brief Title: Hepatitis B Virus Antibody Booster Program for the Production of Hepatitis B Immune Globulin (HBIG)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Prematurely terminated due to failure to meet study objectives.
Sponsor: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HB-012
Record Dates: First submitted 2011-02-25; First posted 2011-03-09 (Estimated); Results first posted 2021-08-17 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Hepatitis B Vaccines; Engerix-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Schedule 1- Standard dose primary vaccination series (Active Comparator): Schedule 1 subjects received 20 µg/1.0 mL of Engerix-B® on Day 0, Day 30, Day 180 with booster of 20 µg/1.0 mL of Engerix-B® every 120 days (4 months) (after Day 180 vaccination)
  Interventions: Biological: hepatitis B vaccine
- Schedule 2 - High dose primary vaccination series (Experimental): Schedule 1 subjects received 40 µg/1.0 mL of Engerix-B® on Day 0, Day 30, Day 60, Day 180 with booster of 20 µg/1.0 mL of Engerix-B® every 120 days (4 months) (after Day 180 vaccination)
  Interventions: Biological: hepatitis B vaccine

INTERVENTIONS:
Biological: hepatitis B vaccine — Primary vaccination series 20 µg/1.0 mL at baseline, month 1, month 6; followed by booster vaccinations 20 µg/1.0 mL
  Other Names: Engerix-B
  Arms: Schedule 1- Standard dose primary vaccination series
Biological: hepatitis B vaccine — Primary vaccination series 40 µg/2.0 mL at baseline, month 1, month 2, month 6; followed by booster vaccinations 20 µg/1.0 mL
  Other Names: Engerix-B
  Arms: Schedule 2 - High dose primary vaccination series

SUMMARY:
Hepatitis B Virus Antibody Booster Program

DETAILED DESCRIPTION:
The purpose of this study is to vaccinate plasmapheresis donors for collection of high titer plasma to be used in the manufacture of Hepatitis B Immune Globulin (HBIG).

ELIGIBILITY:
Inclusion Criteria

* Age 20-55 years.
* Naïve or previously hepatitis B-vaccinated males or females.
* Normal and healthy as determined by medical history, physical exam, vital signs and clinical laboratory tests
* Subject must meet all required/recommended subject suitability criteria that pertain to normal source plasma donors with the following exception:
* Subjects who previously tested positive for HBsAg may be accepted into the anti- HBs program provided they now test negative and meet all other normal donor suitability criteria.
* Written informed consent.

Exclusion Criteria:

* Subjects who have received a hepatitis B vaccination in the previous six months.
* History of hypersensitivity to yeast or any components of the Engerix-B® vaccine
* History of hypersensitivity to any hepatitis B-containing vaccine.
* Use of any investigational product within the past 30 days or during the course of the study.
* Use of steroids or immunosuppressives during the study period.
* Received immunosuppressive therapy (including systemic steroids) within 30 days before study entry
* Subjects who have received cytotoxic therapy (in the previous 5 years prior to study entry)
* Received parenteral immune globulin products or blood products within 3 months before study entry with the following exceptions:
* RhoGAM (or equivalent anti-D immune globulin) within 6 weeks before study entry;
* Pertussis immune globulin: no exclusion
* Received parenteral immune globulin products or blood products (within 3 months before study entry)
* Past, present, or suspected IV drug use
* Positive HIV, HBV* or HCV test result (*except as described above in Inclusion Criteria)
* Autoimmune disease (such as, but not limited to demyelinating disease)
* Subjects with cancer, heart disease (including hospitalization for myocardial infarction, arrhythmia, syncope, congestive heart failure), uncontrolled hypertension, uncontrolled insulin-dependent diabetes mellitus, seizures, kidney disease
* Severely or morbidly obese, or higher obesity classification, which corresponds to BMI of 35 or higher
* Pregnancy or lactation.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03-11 (Actual); Study Completion 2011-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Brown, MD, Principal Investigator — Cangene Corporation; Gerald Winnan, MD, Principal Investigator — Cangene Corporation
Locations (2):
- United States (2):
  - Cangene Plasma Resources, Mid-Florida, Altamonte Springs, Florida
  - Cangene Plasma Resources, Frederick, Frederick, Maryland

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This reporting only covers the interim analysis data collected within a 12 month period between enrolment of the first subject on 9 September 2009 and the interim analysis report cut off date of 1 September 2010 hence the enrollment number being less than the number of participants specified in the protocol.
Groups:
- Schedule 1 - Standard Dose Primary Vaccination Series: hepatitis B vaccine: Primary vaccination series 20 ug/1.0 mL at baseline, month 1, month 6; followed by booster vaccinations 20 ug/1.0 mL every 4 months
- Schedule 2 - High Dose Primary Vaccination Series: hepatitis B vaccine: Primary vaccination series 40 ug/2.0 mL at baseline, month 1, month 2, month 6; followed by booster vaccinations 20 ug/1.0 mL every 4 months
Period: Overall Study
Arm/Group | Schedule 1 - Standard Dose Primary Vaccination Series | Schedule 2 - High Dose Primary Vaccination Series
Started | 72 | 69
Completed | 28 | 29
Not Completed | 44 | 40

BASELINE CHARACTERISTICS:
Groups:
- Schedule 1- Standard Dose Primary Vaccination Series: Schedule 1 subjects will receive 20 µg/1.0 mL of Engerix-B® on Day 0, Day 30, Day 180 with booster of 20 µg/1.0 mL of Engerix-B® every 120 days (4 months) (after Day 180 vaccination)
  hepatitis B vaccine: Primary vaccination series 20 µg/1.0 mL at baseline, month 1, month 6; followed by booster vaccinations 20 µg/1.0 mL
- Schedule 2 - High Dose Primary Vaccination Series: Schedule 2 subjects will receive 40 µg/1.0 mL of Engerix-B® on Day 0, Day 30, Day 60, Day 180 with booster of 20 µg/1.0 mL of Engerix-B® every 120 days (4 months) (after Day 180 vaccination)
  hepatitis B vaccine: Primary vaccination series 40 µg/2.0 mL at baseline, month 1, month 2, month 6; followed by booster vaccinations 20 µg/1.0 mL
- Total: Total of all reporting groups
Arm/Group | Schedule 1- Standard Dose Primary Vaccination Series | Schedule 2 - High Dose Primary Vaccination Series | Total
Number analyzed (Participants) | 72 | 69 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (8.4) | 36.5 (9.5) | 35.5 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 51 | 46 | 97
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 56 | 54 | 110
  Black/African American | 8 | 8 | 16
  Asian | 2 | 1 | 3
  Other | 5 | 5 | 10
  Multiple races | 1 | 1 | 2
Hepatitis B vaccination status at Baseline [Count of Participants; unit: Participants]
  No vaccination previously | 34 | 32 | 66
  Previously vaccinated | 38 | 37 | 75
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.4 (3.6) | 27.7 (3.9) | 27.6 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Comparison Between Vaccination Schedules Using Day 210 Anti-HBs Antibody Titers AUC(0-t)
Description: The primary endpoint for study HB-012 is area under the anti-HBs antibody concentration-time curve (AUC0-t) through Day 210. This endpoint was chosen because it allowed for the assessment of changes in anti HBs antibody concentration over time, and addressed one of the study objectives: to determine the effectiveness of Engerix-B booster vaccinations in the production of high anti-HBs titer plasma. By comparing AUC0-t between the two dosing schedules, the primary endpoint of AUC0-t also addressed the study objective to determine the optimal vaccination schedule to obtain high anti-HBs titer plasma for the manufacture of HepaGam B.
Time Frame: Day 0 to Day 210
Population: The efficacy analysis population was used to assess the primary endpoint and to generate study conclusions. The efficacy analysis population included all subjects who were vaccinated prior to the interim analysis cut-off date of 1 September 2010 and assessed on visit Day 210.
Measure: Mean (Standard Deviation); unit: IU*days/mL
Arm/Group | Schedule 1- Standard Dose Primary Vaccination Series | Schedule 2 - High Dose Primary Vaccination Series
Number analyzed (Participants) | 28 | 29
IU*days/mL | 1675.8 (3065.6) | 4124.8 (1097.3)
Statistical Analysis 1: Comparison: Schedule 1- Standard Dose Primary Vaccination Series vs Schedule 2 - High Dose Primary Vaccination Series; Test type: Superiority; p = 0.96, t-test, 2 sided

2. Secondary Outcome: Comparison Between Vaccination Schedules Using Anti-HBs Titers on Day 210
Description: Anti-HBs titers on Day 210 were assessed as a measure of the anti-HBs level attained following completion of the primary vaccination series; the final primary-series vaccination was administered for both Schedules on Day 180.
Time Frame: Day 210
Population: The population used for this analysis, efficacy population responders, includes any subject who reached Day 210 (with the exception of subjects with all anti-HBs titer results < 2 IU/mL who were considered non-responders), 14 in Schedule 1 and 21 in Schedule 2. However, four subjects (1 in schedule 1 and 3 in schedule 2) were excluded due to missing day 210 titers.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Schedule 1- Standard Dose Primary Vaccination Series | Schedule 2 - High Dose Primary Vaccination Series
Number analyzed (Participants) | 13 | 18
IU/mL | 14.2 (14) | 31.1 (47.3)
Statistical Analysis 1: Comparison: Schedule 1- Standard Dose Primary Vaccination Series vs Schedule 2 - High Dose Primary Vaccination Series; Test type: Superiority; p = 0.36, t-test, 2 sided

3. Secondary Outcome: Comparison Between Vaccination Schedules Using Time to Reach 55 IU/mL Anti-HBs Plasma Titer Level
Description: Time to reach 55 IU/mL was calculated based on the actual time, in days, from the baseline visit (Day 0) to the first time to reach an anti-HBs titer of 55 IU/mL using Kaplan - Meier methods.
Time Frame: up to Day 258
Population: The efficacy population responder subset was used. If a subject's anti-HBs titer levels did not reach 55 IU/mL on or before the cut-off date September 1, 2010, the subject was included as a censored observation. The last anti-HBs assessment date or interim analysis cut-off date, whichever was later, was used as the censoring date. In schedule 1, 3 subjects reached anti-HBs titer level of 55 IU/mL. In schedule 2, 4 subjects reached a titer of 55 IU/mL.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Schedule 2 - High Dose Primary Vaccination Series: Schedule 1 subjects will receive 40 µg/1.0 mL of Engerix-B® on Day 0, Day 30, Day 60, Day 180 with booster of 20 µg/1.0 mL of Engerix-B® every 120 days (4 months) (after Day 180 vaccination)
  hepatitis B vaccine: Primary vaccination series 40 µg/2.0 mL at baseline, month 1, month 2, month 6; followed by booster vaccinations 20 µg/1.0 mL
Arm/Group | Schedule 1- Standard Dose Primary Vaccination Series | Schedule 2 - High Dose Primary Vaccination Series
Number analyzed (Participants) | 14 | 21
Days | NA [133 to NA] — Insufficient number of patients with events. | NA [NA to NA] — Insufficient number of patients with events.
Statistical Analysis 1: Comparison: Schedule 1- Standard Dose Primary Vaccination Series vs Schedule 2 - High Dose Primary Vaccination Series; Test type: Superiority; p = 0.84, Log Rank

4. Secondary Outcome: Time to Reach Anti-HBs Level of 80 IU/mL
Description: Time to reach 80 IU/mL was calculated based on the actual time, in days, from the baseline visit (Day 0) to the first time to reach an anti-HBs titer of 80 IU/mL.
Time Frame: 0-12 months
Population: The efficacy population responder subset was used. If a subject's anti-HBs titer levels did not reach 80 IU/mL on or before the cut-off date September 1, 2010, the subject was included as a censored observation. The last anti-HBs assessment date or interim analysis cut-off date, whichever was later, was used as the censoring date. In schedule 1, no subjects reached anti-HBs titer level of 80 IU/mL. In schedule 2, 2 subjects reached a titer of 80 IU/mL.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Schedule 1- Standard Dose Primary Vaccination Series | Schedule 2 - High Dose Primary Vaccination Series
Number analyzed (Participants) | 14 | 21
Days | NA [NA to NA] — Insufficient number of patients with events. | NA [NA to NA] — Insufficient number of patients with events.
Statistical Analysis 1: Comparison: Schedule 1- Standard Dose Primary Vaccination Series vs Schedule 2 - High Dose Primary Vaccination Series; Test type: Superiority; p = 0.24, Log Rank

5. Secondary Outcome: Comparison Between Vaccination Schedules Using Time to Peak Anti-HBs Titer
Description: Time to reach peak anti-HBs plasma titer was calculated based on the actual times in days, from the baseline visit (Day 0) to the peak titer using Kaplan-Meier methods.
Time Frame: Up to Day 258
Population: The efficacy population responder subset was used. The interim analysis cut-off date was used as the censoring date, except in the case where the subject was lost to follow-up or withdrawn prior to the interim analysis cut off date.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Schedule 1- Standard Dose Primary Vaccination Series | Schedule 2 - High Dose Primary Vaccination Series
Number analyzed (Participants) | 14 | 21
days | 119.2 (88.0) | 153.3 (86.9)
Statistical Analysis 1: Comparison: Schedule 1- Standard Dose Primary Vaccination Series vs Schedule 2 - High Dose Primary Vaccination Series; Test type: Superiority; p = 0.27, Log Rank

ADVERSE EVENTS:
Time Frame: Adverse events were collected for a total of 7 days using diary cards after each vaccination, for the duration of the study until the interim reporting cut off date of 1 September 2010 (approximately 357 days).
Description: Adverse events were elicited by the investigator (or designate) asking the patient non leading questions at each study visit, and at plasmapheresis visits that fall within 7 days of vaccination. Subjects were questioned about SAEs throughout the study.
Arm/Group | Schedule 1- Standard Dose Primary Vaccination Series | Schedule 2 - High Dose Primary Vaccination Series
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/69
Serious Adverse Events (participants affected / at risk) | 1/72 | 0/69
Other Adverse Events (participants affected / at risk) | 25/72 | 37/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Schedule 1- Standard Dose Primary Vaccination Series (N=72) | Schedule 2 - High Dose Primary Vaccination Series (N=69)
Hepatomegaly and elevated liver enzymes (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Schedule 1- Standard Dose Primary Vaccination Series (N=72) | Schedule 2 - High Dose Primary Vaccination Series (N=69)
EOSINOPHILIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
HYPOCHROMIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
CERUMEN IMPACTION (Ear and labyrinth disorders) | 0 (0) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 1 (2)
CHEST DISCOMFORT (General disorders) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 1 (1)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 1 (1)
INJECTION SITE INFLAMMATION (General disorders) | 0 (0) | 2 (2)
INJECTION SITE PAIN (General disorders) | 9 (12) | 12 (19)
PYREXIA (General disorders) | 1 (1) | 0 (0)
HEPATITIS (Hepatobiliary disorders) | 2 (2) | 0 (0)
ALLERGY TO ANIMAL (Immune system disorders) | 0 (0) | 1 (1)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 3 (3)
MULTIPLE ALLERGIES (Immune system disorders) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 1 (1)
INFLUENZA (Infections and infestations) | 1 (1) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 1 (1)
OTITIS EXTERNA (Infections and infestations) | 1 (1) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
VIRAEMIA (Infections and infestations) | 1 (1) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 3 (3) | 2 (2)
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
LIMB INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
BLOOD GLUCOSE DECREASED (Investigations) | 0 (0) | 2 (2)
BLOOD GLUCOSE INCREASED (Investigations) | 1 (1) | 2 (2)
CARBON DIOXIDE DECREASED (Investigations) | 0 (0) | 1 (1)
EOSINOPHIL COUNT INCREASED (Investigations) | 0 (0) | 1 (2)
HEPATITIS B SURFACE ANTIGEN POSITIVE (Investigations) | 0 (0) | 1 (1)
HIV TEST NEGATIVE (Investigations) | 0 (0) | 1 (1)
NEUTROPHIL COUNT INCREASED (Investigations) | 0 (0) | 1 (1)
TREPONEMA TEST FALSE POSITIVE (Investigations) | 0 (0) | 1 (1)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 (0) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
HEADACHE (Nervous system disorders) | 5 (7) | 9 (11)
MIGRAINE (Nervous system disorders) | 1 (1) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
SINUS HEADACHE (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 2 (2)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (2) | 0 (0)
STRESS (Psychiatric disorders) | 1 (1) | 0 (0)
CHROMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
URINARY TRACT PAIN (Renal and urinary disorders) | 0 (0) | 1 (1)
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This reporting only covers the interim analysis data collected within a 12 month period between enrolment of the first subject on 9 September 2009 and the interim analysis report cut off date of 1 September 2010.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No